CLINICAL TRIAL: NCT06728995
Title: Prediction of Recipient Renal Function in Living Donor Kidney Transplantation Using Baseline Characteristics and Donor Renal Volume
Brief Title: Renal Function Prediction in Living Donor Transplant Using Baseline Data
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang-Il Min, MD, PhD, Professor, Seoul National University Hospital
Other Study IDs: SNUH-Volumetry_KT Recipient; H-2205-051-1322 (Other: Seoul National University Hospital Institutional Review Board)
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Renal Transplanted Recipients; Kidney Function
Keywords: renal transplantation; kidney volume; predictive model; machine learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: All participants included in the retrospective study who underwent living-donor kidney transplantation. No interventions were applied as this is an observational study.

SUMMARY:
This study aims to predict early post-transplant kidney function in living donor kidney transplant recipients using baseline characteristics of donors and recipients. The study involves analyzing pre-transplant data to develop a machine learning model that predicts serum creatinine levels one year post-transplant. This research may improve decision-making and outcomes for transplant patients

ELIGIBILITY:
Inclusion Criteria:

- Recipients and donors of living-donor kidney transplantation.

Exclusion Criteria:

* Donors or recipients with follow-up durations of less than 1 year.
* Recipients who received simultaneous organ transplantation in addition to kidney transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited from Seoul National University Hospital, Severance Hospital, and Bundang Seoul National University Hospital, encompassing recipients and donors involved in living-donor kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Lowest Serum Creatinine Level | Within one year post-transplant.
  Measurement of the lowest serum creatinine level post-transplant to evaluate kidney function.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to researchers upon reasonable request, subject to approval by the IRB

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT06728995/Prot_SAP_000.pdf